CLINICAL TRIAL: NCT06006403
Title: Clinical Study of Targeting CD123 Chimeric Antigen Receptor Natural Killer Cells (CAR-NK) in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm
Brief Title: Safety and Efficacy of CD123-targeted CAR-NK for Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC050
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia; Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN); Relapse Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Myeloid Leukemia (Experimental): Infusion of CD123-targeted CAR-NK cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CD123 targeted CAR-NK cells
- Blastic Plasmacytoid Dendritic Cell Neoplasm (Experimental): Infusion of CD123-targeted CAR-NK cells by dose of 1-10x10^6 cells/kg
  Interventions: Biological: CD123 targeted CAR-NK cells

INTERVENTIONS:
Biological: CD123 targeted CAR-NK cells — Administration method: intravenous infusion； Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This study is a single-arm, open-label, dose-escalating + dose-expansion clinical study, aiming to evaluate the safety and efficacy of targeting CD123 CAR-NK cell preparations in Relapsed/refractory acute myeloid leukemia (AML) or blastocytic plasmacytoid dendritic cell neoplasm (BPDCN). The pharmacokinetic characteristics of CAR-NK cell preparations for the treatment of patients with Relapsed/refractory acute myeloid leukemia or blastocytic plasmacytoid dendritic cell neoplasm were obtained and the recommended dose.

DETAILED DESCRIPTION:
According to the different disease type, it is divided into two subgroups: AML and BPDCN. Each subgroup includes a dose exploration stage (Part A) and a dose expansion stage (Part B). 3 patients were explored, starting from the low-dose group, and in the dose expansion phase, the safety and efficacy were further verified according to the safe recommended dose obtained in the dose exploration phase.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited, age 18-75 years old (including the threshold value);
2. The expression of CD123 in tumor cells was detected by flow cytometry.
3. Patients with relapsed/refractory AML or BPDCN diagnosed with CD123 positive: 1) AML: a. Recurrent: After complete response (CR), the recurrence of leukemia cells in peripheral blood or bone marrow original cells ≥5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or the occurrence of extramedullary leukemia cell infiltration; b. Refractory: refers to those who have failed to receive 2 courses of treatment with standard protocols; Patients recurrence within 12 months after CR with consolidation and intensive treatment; Recurrence after 12 months but failed to respond to conventional chemotherapy; 2 or more relapses; Extramedullary leukemia persists;

2) BPDCN: has failed to receive guidelines-recommended salvage therapy or is unable to tolerate current therapy, and has persistent or recurrent disease in any of the peripheral blood, bone marrow, lymph nodes, spleen, skin lesions, or other site lesions.

4. Expected survival time is more than 12 weeks;

5. ECOG 0-2 points (Appendix 2);

6. No serious mental disorders; The functions of important organs are basically normal:

1. Cardiac function: echocardiography indicated cardiac ejection fraction ≥50%, and no obvious abnormality was found in electrocardiogram;
2. Renal function: serum creatinine ≤2.0×ULN;
3. Liver function: ALT and AST ≤ 3.0×ULN;
4. Total bilirubin and alkaline phosphatase ≤ 2.0×ULN (Gilbert syndrome ≤ 3.0×ULN);
5. Blood oxygen saturation > 92%.

   7. The patient or his/her guardian agrees to participate in the clinical trial and signs the ICF, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Prior to screening, the following anti-tumor therapies were received: chemotherapy, targeted therapy, or other investigational drug treatment within 14 days or at least 5 half-lives (whichever is shorter), except in cases where disease progression has been confirmed after treatment;
2. had a cerebrovascular accident or seizure within 6 months before signing the ICF;
3. There is an active or uncontrolled infection that requires systemic treatment within 1 week prior to screening;
4. suffering from any of the following heart diseases:

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. Had myocardial infarction or coronary artery bypass grafting (CABG) within ≤6 months before enrollment;
   3. A history of clinically significant ventricular arrhythmia, or unexplained syncope (other than those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
5. combined with active hepatitis B;
6. Combined with active autoimmune diseases, long-term immunosuppressive therapy is required;
7. have other malignancies, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
8. Had received live attenuated vaccine within 4 weeks prior to screening;
9. Women who are pregnant or breastfeeding, and male or female subjects who plan to have a family within 1 year after receiving CAR T cell transfusion;
10. Circumstances deemed unsuitable for participation in the study by other researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-NK cell preparations in the treatment of Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm[Safety and Tolerability] | 1 month
  The incidence of adverse events after CD123 CAR-NK cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)
To evaluate the efficacy of CAR-NK cell preparations in the treatment of Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm[Effectiveness] | 1month,3months
  Objective response rate at 4W±7D and 3M±7D after CAR-NK infusion (Objective response rate includes CR, CRi)

SECONDARY OUTCOMES:
AUCS of CD123 CAR-NK cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of CD123 CAR-NK cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of CEA CAR-T cells expanded in peripheral blood
TMAX of CD123 CAR-NK cells[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of CD123 CAR-NK cells[Cell dynamics] | 3 months
  The degree of clearance of malignant cells in peripheral blood was detected by blood smear at each time point，and the concentration level of serum cytoplasmic factors such as CRP and IL-6 were detected by ELISA at each time point

OTHER OUTCOMES:
Duration of Response (DOR) of CD123 CAR-NK treatment in patients with Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm[Effectiveness] | 2 years
  DOR will be assessed from the first assessment of CR/CRi to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CD123 CAR-NK treatment in patients with Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm[Effectiveness] | 2 years
  PFS will be assessed from the first CD123 CAR-NK cell infusion to death from any cause or the first assessment of progression
Overall survival(OS)of CD123 CAR-NK treatment in patients with Relapsed/Refractory Acute Myeloid Leukemia or Blastic Plasmacytoid Dendritic Cell Neoplasm[Effectiveness] | 2 years
  OS will be assessed from the first CD123 CAR-NK cell infusion to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wei, M.D, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China